CLINICAL TRIAL: NCT01625156
Title: A Phase 1 Study of ARQ 197 in Combination With Temsirolimus in Advanced Solid Tumors
Brief Title: Tivantinib and Temsirolimus in Treating Patients With Solid Tumors That is Metastatic or Cannot be Removed by Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-00949; NCI-2012-00949 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI 9145; 905854-02-06; NCI-2012-00974; CO 11914 (Other: University of Wisconsin Hospital and Clinics); 9145 (Other: CTEP); P30CA014520 (NIH); U01CA062491 (NIH)
Record Dates: First submitted 2012-06-18; First posted 2012-06-21 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-05

CONDITIONS: Adult Solid Neoplasm
MeSH Terms: interventions — temsirolimus; Sirolimus; ARQ 197

ARMS (1):
- Treatment (tivantinib, temsirolimus) (Experimental): Patients receive tivantinib PO BID and temsirolimus IV over 30 minutes on days 1, 8, 15, and 22 (days 8, 15, 22, and 29 of course 1). Courses repeat every 28 days (35 days in course 1) in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Temsirolimus; Drug: Tivantinib

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Temsirolimus — Given IV
  Other Names: CCI-779; CCI-779 Rapamycin Analog; Cell Cycle Inhibitor 779; Rapamycin Analog; Rapamycin Analog CCI-779; Torisel
Drug: Tivantinib — Given PO
  Other Names: ARQ 197; ARQ-197; c-Met Inhibitor ARQ 197

SUMMARY:
This phase I trial studies the side effects and best dose of tivantinib when given in combination with temsirolimus in treating patients with solid tumors that have spread to other parts of the body or cannot be removed by surgery. Tivantinib and temsirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of ARQ197 (tivantinib) in combination with temsirolimus in adult subjects with advanced solid tumors who are extensive cytochrome P450, family 2, subfamily C, polypeptide 19 (CYP2C19) metabolizers.

SECONDARY OBJECTIVES:

I. To characterize the tolerability and/or MTD of ARQ 197 and in combination with temsirolimus in adult subjects who are poor CYP2C19 metabolizers (CYP2C19*2/*2, *2/*3 or *3/*3 polymorphisms).

II. To identify the pharmacokinetic parameters of ARQ 197 after a single dose and at steady state in extensive and poor CYP2C19 metabolizers.

III. To assess the steady state pharmacokinetics of ARQ 197 alone and in combination with temsirolimus.

IV. To determine impact of cytochrome P450, family 3, subfamily A, polypeptide 4/cytochrome P450, family 3, subfamily A, polypeptide 5 (CYP3A4/5) polymorphisms on ARQ 197 pharmacokinetic parameters.

V. To determine the pharmacokinetics of temsirolimus and its active metabolite sirolimus in combination with ARQ 197 and compare to historical pharmacokinetic data.

VI. To determine impact of CYP3A4/5 polymorphisms on temsirolimus pharmacokinetic parameters.

VII. To describe the dose-limiting toxicities and determine the safety profile of the combination of ARQ 197 and temsirolimus.

VIII. To evaluate the preliminary anti-tumor activity of ARQ197 and temsirolimus in patients with advanced solid tumors.

IX. To correlate archived tumor tissue expression of c-Met with objective response to ARQ 197 and temsirolimus therapy.

OUTLINE: This is a dose-escalation study of tivantinib.

Patients receive tivantinib orally (PO) twice daily (BID) and temsirolimus intravenously (IV) over 30 minutes on days 1, 8, 15, and 22 (days 8, 15, 22, and 29 of course 1). Courses repeat every 28 days (35 days in course 1) in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for at least 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed solid malignancy (excluding lymphoma) that is metastatic or unresectable and for which standard curative or palliative systemic therapies (such as chemotherapy, targeted therapies or immunotherapy) do not exist or are no longer effective
* Patients must have measurable or evaluable disease, as defined by Response Evaluation Criteria In Solid Tumors (RECIST) 1.1
* No prior treatment with temsirolimus or an agent specifically targeting met proto-oncogene (c-Met)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 12 weeks
* Hemoglobin >= 9.0 g/dL
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 X institutional upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< institutional upper limit of normal
* Serum creatinine =< institutional upper limit of normal or creatinine clearance (either estimated or calculated) >= 60 mL/min/1.73 m for patients with creatinine levels above institutional normal
* Fasting glucose =< 150 mg/dL
* Fasting cholesterol level < 350 mg/dl
* Fasting triglycerides =< 300 mg/dl
* Phosphorus >= institutional lower limit of normal (repletion allowed)
* Patients with treated, stable brain metastases are allowed to enroll; patients must be at least 4 weeks from radiation and off any medications used to treat brain metastases including steroids; patients are allowed to be on antiepileptic medications that are not metabolized by cytochrome P450 3A4 or 2C19; patients with brain metastases must have stable brain imaging within 4 weeks prior to starting study
* Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and up to 3 months after discontinuation of study drugs; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of ARQ 197 administration; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Any of the following:

  * Chemotherapy =< 3 weeks prior to entering the study (6 weeks for nitrosoureas or mitomycin C)
  * Radiotherapy, endocrine therapy or targeted therapy for malignancy =< 2 weeks prior to registration
  * Patients who have not recovered (=< grade 1) from adverse events due to agents administered more than 4 weeks earlier (tolerable grade 2 adverse events may be allowed at the discretion of the investigator; diarrhea must be grade 1 or lower without the scheduled use of antidiarrheal medications)
  * Prior anticancer therapy with an mammalian target of rapamycin (mTOR) inhibitor (everolimus, temsirolimus, desferolimus) or agent specifically targeting c-Met
* Patients who are receiving any other investigational agents
* Patients may not have clinically symptomatic hypothyroidism; testing is not required for eligibility
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ARQ 197 or temsirolimus
* ARQ 197 is a sensitive substrate for 2C19 and 3A4, a strong inhibitor for 2C19 and moderate inhibitor by in vitro data only for 3A4; temsirolimus is a sensitive substrate for CYP 3A4 and a weak inhibitor of CYP2D6 and CYP3A4/5; per the UWinRx Drug Interaction Policy, the following medications are contraindicated or must be used with caution
* Contraindicated:

  * CYP2C19 sensitive substrates (unless close monitoring with labs or drug levels with dose adjustments is feasible), inducers, and moderate/strong inhibitors of CYP2C19; patients taking these concurrent medications are ineligible unless they can be switched to alternative medications prior to initiation of the study
  * CYP3A4/5 inducers and moderate/strong inhibitors of CYP3A4/5; patients taking these concurrent medications are ineligible unless they can be switched to alternative medications prior to initiation of the study
* Use with caution:

  * CYP2C19 non-sensitive substrates with a narrow therapeutic window and weak inhibitors are permitted if no acceptable alternatives are available as determined by the treating physician; however, caution should be used; consider monitoring with labs or drug levels and dose adjustments of the medication if feasible; other non-sensitive substrates are allowed on study
  * CYP3A4/5 sensitive substrates and any non-sensitive substrates with a narrow therapeutic window and weak inhibitors are permitted if no acceptable alternatives are available as determined by the treating physician; however, caution should be used; consider monitoring with labs or drug levels and dose adjustments of the medication if feasible; other non-sensitive substrates are allowed on study
  * CYP2D6 inducers, moderate/strong inhibitors or sensitive substrates are permitted if no acceptable alternatives are available; however, caution should be used; other non-sensitive substrates or weak inhibitors of CYP2D6 are allowed on study
* History of congestive heart failure defined as class II to IV per New York Heart Association (NYHA) classification; active coronary artery disease (CAD); clinically significant bradycardia (< 50 beats per minute [bpm]) or other uncontrolled, cardiac arrhythmia defined as >= grade 3 according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.0, or uncontrolled hypertension (as determined by the investigator); myocardial infarction occurring within 6 months prior to study entry (myocardial infarction occurring > 6 months prior to study entry is permitted)
* Patients with uncontrolled diabetes (as determined by the investigator); well-controlled diabetic patients with fasting glucose < 150 are eligible if they have been on stable doses of medications for diabetes for at least 4 weeks prior to study entry
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded; breastfeeding should be discontinued if the mother is treated on this study
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Patients with malabsorption syndrome or other condition that would interfere with intestinal absorption of pills; patients must be able to swallow pills

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-05; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
MTD and RP2D of tivantinib in combination with temsirolimus defined as the highest safely tolerated dose where 0/6 or 1/6 patients experience a dose-limiting toxicity (DLT) and two or more patients have experienced a DLT at the next higher dose level | First 35 days
  Categorized according to NCI Common Toxicity Criteria version 4.0.

SECONDARY OUTCOMES:
Incidence of adverse events and toxicities of tivantinib in combination with temsirolimus | Up to 4 weeks after completion of study treatment
  Categorized according to NCI Common Toxicity Criteria version 4.0. Summarized in terms of type, severity (grade 1-5), and dose level in tabular format. Wilson score method will be used to construct confidence intervals.
Pharmacokinetic analysis | Pre-dose, 0.5, 1, 2, 4, 8, and 12 hours (days 1 and 7), pre-dose and 0.5 hours (day 8), pre-dose (days 15 and 22 of course 1 and day 1 of course 2)
  Plots of individual, mean, and median plasma concentration versus time will be presented where appropriate. The comparison of PK parameters between dose levels will be performed using a two-sample t-test.
Response rate validated by the RECIST criteria | Up to 4 weeks after completion of study treatment
  Summarized by simple descriptive summary statistics delineating complete and partial responses as well as stable and progressive disease. Ninety-five percent confidence intervals will be constructed using the Wilson Score method.

OTHER OUTCOMES:
Tumor tissue expression levels of c-Met | Up to course 2, day 1
  Tumor tissue expression levels of c-Met will be summarized using standard descriptive statistics (for patients in the dose expansion cohort). A two-sample t-test will be used to compare mean tumor expression levels of c-Met between responders (complete response [CR] or partial response [PR]) versus non-responders (stable disease [SD], progressive disease), and between patients with clinical benefit (CR, PR or SD) versus patients with progressive disease.

CONTACTS AND LOCATIONS:
Overall Officials: Kari Wisinski, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Wisconsin Clinical Cancer Center, Milwaukee, Wisconsin